CLINICAL TRIAL: NCT01700400
Title: Phase I Dose Escalation Study of Everolimus, Pemetrexed, Carboplatin, and Bevacizumab in Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Study of Everolimus, Pemetrexed, Carboplatin, and Bevacizumab to Treat Stage IV Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research and Biostatistics Clinical Trials Consortium (Network)
Collaborators: University of Arizona (Other); Providence Cancer Center, Earle A. Chiles Research Institute (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAB CTC 10-001
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Non Small Cell Lung Cancer; Advanced Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Everolimus; Pemetrexed; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Phase I Dose Escalation (Experimental): Pemetrexed: intravenous; 500 mg/m² for Dose Levels 1, 2 and 3
  Carboplatin: intravenous; 5 AUC for Dose Level 1; 6 AUC for Dose Levels 2 and 3
  Bevacizumab: intravenous; 15 mg/kg for Dose Levels 1, 2, and 3
  Everolimus: oral, 2.5 mg/day for Dose Levels 1 and 2; 5.0 mg/day for Dose Level 3
  Interventions: Drug: Everolimus; Drug: Pemetrexed; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Everolimus
  Other Names: Afinitor; Zortress; RAD001
Drug: Pemetrexed
  Other Names: Alimta
Drug: Carboplatin
  Other Names: Paraplatin; CBDCA
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine whether the investigational study drug everolimus may be used to increase the effectiveness of chemotherapy treatment for patients with advanced lung cancer.

DETAILED DESCRIPTION:
Advanced lung cancer remains an incurable disease although new agents and new treatment strategies have resulted in improved survival outcomes for patients. Most recently there has been interest in augmenting tumor response to chemotherapy by the addition of drugs which inhibit tumor cell growth and proliferation. Everolimus is a new cancer drug which works as an inhibitor of mammalian target of rapamycin (or mTOR), mTOR is a protein that is part of a signaling pathway which can cause cancer cells to divide. Everolimus when used alone as a single agent has produced some response as well as prolonged stable disease in both chemo-naïve and pre-treated non-small cell lung cancer. The goal of this study is to evaluate the safety of everolimus with combined other cancer drugs called pemetrexed, carboplatin, and bevacizumab. Pemetrexed and carboplatin are both chemotherapy drugs and bevacizumab inhibits the growth of new blood vessels.

Patients will be entered onto dosing cohorts of 3 patients according to the following dose escalation scheme. The first cohort will begin at dose level 1. At least three patients on each dose level must have completed cycle one before the study leadership (principal investigators, study statisticians) will allow patients to be enrolled onto the successive dose level.

Dose Levels: 1, 2, 3

Pemetrexed (mg/m²): 500, 500, 500

Carboplatin (AUC): 5, 6, 6

Bevacizumab (mg/kg): 15, 15, 15

Everolimus (mg/day): 2.5, 2.5, 5.0

The purpose of this study is to determine the maximum tolerated dose, or MTD, for the combination of everolimus with pemetrexed, carboplatin, and bevacizumab in patients with Stage IV non-squamous, non small cell lung cancer.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Signed informed consent
   2. Confirmed diagnosis of Stage IV non-squamous non-small cell lung cancer
   3. CT of the chest, abdomen, and pelvis which shows metastatic disease. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
   4. At least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
   5. Age ≥ 18 years
   6. Normal blood function levels as evidenced by laboratory tests.
   7. Adequate liver, kidney and blood chemistry function.
   8. Adequate blood clotting levels
   9. Urine dipstick levels of protein must be between 0-1+.
   10. Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x IULN. Testing must be performed within 14 days prior to enrollment.
   11. The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed.
   12. No prior treatment with everolimus. Prior treatment with pemetrexed or carboplatin is allowed, provided no disease progression with prior exposure to drugs. Prior treatment with bevacizumab allowed.
2. Exclusion Criteria:

   1. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
   2. Clinically significant cardiac event such as Myocardial infarction
   3. Inadequately controlled high blood pressure
   4. Active gastrointestinal disease resulting in an inability to take oral or enteral medication via a feeding tube or a requirement for IVplacement; prior surgical procedures affecting absorption; or active peptic ulcer disease
   5. Presence of fluid accumulation which cannot be controlled by drainage
   6. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to enrollment
   7. History of stroke within 6 months prior to enrollment
   8. History of significant vascular disease within 6 months prior to enrollment(i.e., aortic aneurysm)
   9. No unusual bleeding or inability to clot (assuming not on anti-coagulation); patients with a history of DVT and/pr pulmonary embolism are excluded
   10. Serious non-healing wound, ulcer, or bone fracture
   11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, or anticipation of need for major surgical procedure during the course of the study. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
   12. Untreated brain metastases Radiation treatment than 28 days prior to registration. Side effects due to radiation therapy must have resolved.
   13. Coughing up of blood
   14. Excessive protein in your urine
   15. Abnormal levels of lipids in your blood
   16. Previous or current malignancies within the last 3 years, with the exception of cervical cancer and adequately treated basal cell or squamous cell carcinoma of the skin
   17. Prior treatment with any investigational drug within the preceding 4 weeks prior to enrollment
   18. Patients receiving chronic, systemic treatment with corticosteroids or another immunotherapy. Topical or inhaled corticosteroids are allowed.
   19. Patients must not receive immunization with attenuated live vaccines within one week prior to study enrollment or during study period.
   20. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation.
   21. HIV positive
   22. Impairment of stomach or intestinal function or stomach or intestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
   23. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus.
   24. Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus)
   25. Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Define the Maximum Tolerated Dose (MTD) and Recommended Phase Two Dose (RPTD) of the combination of everolimus with pemetrexed, carboplatin, and bevacizumab in patients with Stage IV non-squamous NSCLC. | up to 2 years
  Pemetrexed, carboplatin and bevacizumab will be given intravenously on day 1 of a 21-day cycle with doses determined by the dose level to which the patient is assigned.
  Everolimus will be taken orally days 1-21 of a 21-day cycle. There will be no rest between each 21 day cycle. Tumor scans will be done every 2 treatment cycles. Patients who are not progressing and who are tolerating therapy will be treated with 6 cycles of Pem/Carbo/Bev/Everolimus followed by maintenance Pem/Bev/Everolimus, which will be continued if there is no tumor progression and the patient is tolerating therapy. If there is toxicity related specifically to one of the maintenance drugs, that drug will be discontinued and the other drugs will be maintained.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 2 years
  Dose Limiting Toxicity (DLT) adverse events related to everolimus/pemetrexed/carboplatin/bevacizumab administration in patients with Stage IV non-squamous NSCLC. DLTs will be defined during cycle 1 only. Grading of adverse events will be according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
  Hematologic Adverse Events are defined as:
  Grade 4 neutropenia lasting greater than 5 days; Grade 3 or 4 febrile neutropenia; and/or Grade 4 thrombocytopenia
  Non-hematologic Adverse Events are defined as:
  Grade 3 or greater non-hematologic excluding the following:
  Hypersensitivity reaction grade 3 or 4 occurring on day 1 or day 15; Nausea/vomiting grade 3 or 4 in the absence of optimal antiemetics; Diarrhea grade 3 or 4 in the absence of optimal anti-diarrheal therapy; Asthenia grade 3 or 4 of less than 2 weeks duration; and/or Hyperglycemia grade 3 or 4 temporally related to corticosteroid pre-or post-medication
Antitumor efficacy associated with administration of everolimus/pemetrexed/carboplatin/bevacizumab administration in patients with Stage IV non-squamous NSCLC. | up to 2 years
  number of patients with a response according to the Response Evaluation Criteria in Solid Tumors (RECIST)
Progression-free survival (PFS) | up to 2 years
  time from start of treatment to time of progression or death (overall PFS)
Overall Survival (OS) | up to 2 years
  measured from the start of treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Linda L. Garland, MD, Principal Investigator — University of Arizona; John Crowley, PhD, Study Chair — Cancer Research And Bioststistics
Locations (4):
- United States (4):
  - University of Arizona Cancer Center, Tuscon, Arizona
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Providence Cancer Center, Portland, Oregon
  - Cancer Research And Biostatistics Clinical Trials Consortium, Seattle, Washington

REFERENCES:
- See also: Providence Cancer Center of Portland, Oregon — http://oregon.providence.org/patients/programs/providence-cancer-center/Pages/default.aspx